CLINICAL TRIAL: NCT02603120
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Switching From a Regimen of Dolutegravir and ABC/3TC, or a Fixed Dose Combination (FDC) of ABC/DTG/3TC to a FDC of GS-9883/F/TAF in HIV-1 Infected Subjects Who Are Virologically Suppressed
Brief Title: Safety and Efficacy of Switching From Dolutegravir and ABC/3TC or ABC/DTG/3TC to B/F/TAF in HIV-1 Infected Adults Who Are Virologically Suppressed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-380-1844; 2015-004025-14 (EudraCT Number)
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — abacavir, dolutegravir, and lamivudine drug combination; bictegravir; tenofovir alafenamide; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Blinded Phase: B/F/TAF (Experimental): B/F/TAF + ABC/DTG/3TC placebo for at least 48 weeks
  Interventions: Drug: B/F/TAF; Drug: ABC/DTG/3TC Placebo
- Blinded Phase: ABC/DTG/3TC (Active Comparator): ABC/DTG/3TC + B/F/TAF placebo for at least 48 weeks
  Interventions: Drug: ABC/DTG/3TC; Drug: B/F/TAF Placebo
- Open-Label Phase (Experimental): At the End of Blinded Treatment Visit, if safety and efficacy of B/F/TAF is demonstrated following review of unblinded data, participants in a country where B/F/TAF FDC is not available will be given the option to receive B/F/TAF FDC in an open-label extension phase for up to 96 weeks, or until the product becomes accessible to subjects through an access program, or until Gilead Sciences elects to discontinue the study in that country, whichever occurs first.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: ABC/DTG/3TC — 600/50/300 mg FDC tablets administered orally once daily without regard to food
  Other Names: Triumeq®
  Arms: Blinded Phase: ABC/DTG/3TC
Drug: B/F/TAF — 50/200/25 mg FDC tablets administered orally once daily without regard to food
  Other Names: Bictegravir (previously referred to as GS-9883)/Emtricitabine/Tenofovir Alafenamide; Biktarvy® [BVY]
  Arms: Blinded Phase: B/F/TAF; Open-Label Phase
Drug: ABC/DTG/3TC Placebo — Tablets administered orally once daily without regard to food
  Arms: Blinded Phase: B/F/TAF
Drug: B/F/TAF Placebo — Tablets administered orally once daily without regard to food
  Arms: Blinded Phase: ABC/DTG/3TC

SUMMARY:
The primary objective of this study is to evaluate the efficacy of switching from a regimen of dolutegravir (DTG) and abacavir/lamivudine (ABC/3TC) or a fixed dose combination (FDC) of abacavir/dolutegravir/lamivudine (ABC/DTG/3TC) to a FDC of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) versus continuing DTG and ABC/3TC as the FDC ABC/DTG/3TC in virologically suppressed Human Immunodeficiency Virus- 1 (HIV-1) infected adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Estimated glomerular filtration rate ≥ 50 mL/min (≥ 0.83 mL/sec).
* Currently receiving an antiretroviral regimen of DTG + ABC/3TC, or ABC/DTG/3TC FDC for ≥ 3 months prior to the screening visit.
* HIV ribonucleic acid (RNA) < 50 copies/mL at the screening visit.
* Currently on a stable regimen for ≥ 3 months preceding the screening visit with documented plasma HIV-1 RNA < 50 copies/mL for ≥ 3 months preceding the screening visit (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL).
* Have no documented or suspected resistance to emtricitabine (FTC), tenofovir (TFV), DTG, ABC or 3TC.

Key Exclusion Criteria:

* Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance.
* Active tuberculosis infection.
* Individuals experiencing decompensated cirrhosis (eg, ascites, encephalopathy, or variceal bleeding).
* Females who are pregnant.
* Females who are breastfeeding.
* Acute hepatitis in the 30 days prior to study entry.
* Chronic Hepatitis B Virus (HBV) infection.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (76):
- United States (51):
  - Phoenix, Arizona
  - Beverly Hills, California
  - Los Angeles, California
  - Oakland, California
  - Palm Springs, California
  - Sacramento, California
  - San Leandro, California
  - Washington D.C., District of Columbia
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Ft. Pierce, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Wilton Manors, Florida
  - Augusta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Savannah, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Berkley, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Newark, New Jersey
  - Santa Fe, New Mexico
  - Buffalo, New York
  - New York, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Huntersville, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Longview, Texas
  - Seattle, Washington
  - Spokane, Washington
- Sydney, New South Wales, Australia
- Ghent, Belgium
- Canada (3):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Montreal, Quebec
- France (3):
  - Nantes
  - Nice
  - Paris
- Germany (7):
  - Berlin
  - Bonn
  - Essen
  - Frankfurt am Main
  - Hamburg
  - Munich
  - München
- Roma, Italy
- San Juan, Puerto Rico
- Spain (6):
  - Badalona
  - Barcelona
  - Córdoba
  - Madrid
  - Santiago de Compostela
  - Seville
- United Kingdom (2):
  - Brighton
  - Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Andreatta K, Willkom M, Martin R, Chang S, Wei L, Liu H, Liu YP, Graham H, Quirk E, Martin H, White KL. Switching to bictegravir/emtricitabine/tenofovir alafenamide maintained HIV-1 RNA suppression in participants with archived antiretroviral resistance including M184V/I. J Antimicrob Chemother. 2019 Dec 1;74(12):3555-3564. doi: 10.1093/jac/dkz347. PMID 31430369
- [Result] Molina JM, Ward D, Brar I, Mills A, Stellbrink HJ, Lopez-Cortes L, Ruane P, Podzamczer D, Brinson C, Custodio J, Liu H, Andreatta K, Martin H, Cheng A, Quirk E. Switching to fixed-dose bictegravir, emtricitabine, and tenofovir alafenamide from dolutegravir plus abacavir and lamivudine in virologically suppressed adults with HIV-1: 48 week results of a randomised, double-blind, multicentre, active-controlled, phase 3, non-inferiority trial. Lancet HIV. 2018 Jul;5(7):e357-e365. doi: 10.1016/S2352-3018(18)30092-4. Epub 2018 Jun 18. PMID 29925489
- [Derived] Brar I, Ruane PJ, Berhe M, Brinson C, Benson P, Henry K, Liu H, Andreatta K, Hindman JT, Ramgopal M. Efficacy and safety of switch to bictegravir/emtricitabine/tenofovir alafenamide from dolutegravir/abacavir/lamivudine: Results from an open-label extension of a phase 3 randomized, double-blind, multicenter, active-controlled, non-inferiority study. Medicine (Baltimore). 2025 Feb 21;104(8):e41482. doi: 10.1097/MD.0000000000041482. PMID 39993074
- [Derived] Avihingsanon A, Chetchotisakd P, Kiertiburanakul S, Ratanasuwan W, Siripassorn K, Supparatpinyo K, Martin H, Wang H, Wong T, Wang HY. Efficacy and safety of switching to bictegravir, emtricitabine, and tenofovir alafenamide in virologically suppressed Asian adults living with HIV: A pooled analysis from three international phase III randomized trials. HIV Med. 2023 Mar;24(3):290-300. doi: 10.1111/hiv.13386. Epub 2022 Aug 17. PMID 36912172
- [Derived] Wohl D, Clarke A, Maggiolo F, Garner W, Laouri M, Martin H, Quirk E. Patient-Reported Symptoms Over 48 Weeks Among Participants in Randomized, Double-Blind, Phase III Non-inferiority Trials of Adults with HIV on Co-formulated Bictegravir, Emtricitabine, and Tenofovir Alafenamide versus Co-formulated Abacavir, Dolutegravir, and Lamivudine. Patient. 2018 Oct;11(5):561-573. doi: 10.1007/s40271-018-0322-8. PMID 29956087

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Australia. The first participant was screened on 11 November 2015. The last study visit occurred on 23 October 2019.
Pre-assignment Details: 646 participants were screened.
Groups:
- B/F/TAF: Double-Blind Phase: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) 50/200/25 mg fixed dose combination (FDC) tablet + abacavir/dolutegravir/lamivudine (ABC/DTG/3TC) placebo orally once daily for at least 48 weeks, without regard to food.
  Open-label (OL) Extension Phase: After Week 48, participants in a country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
- ABC/DTG/3TC: Double-Blind Phase: ABC/DTG/3TC (600/50/300 mg) FDC tablet + B/F/TAF placebo orally once daily for at least 48 weeks, without regard to food.
  OL Extension Phase: After Week 48, participants in a country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
Period: Double-Blind Treatment Phase
Arm/Group | B/F/TAF | ABC/DTG/3TC
Started | 284 | 283
Completed | 265 | 267
Not Completed | 19 | 16
Not completed — Withdrew consent | 4 | 8
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 4 | 2
Not completed — Death | 2 | 0
Not completed — Investigator's discretion | 2 | 0
Not completed — Pregnancy | 1 | 1
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Did not receive study drug | 2 | 2
Period: OL Extension B/F/TAF Treatment Phase
Arm/Group | B/F/TAF | ABC/DTG/3TC
Started | 259 | 265
Completed | 254 | 254
Not Completed | 5 | 11
Not completed — Lost to Follow-up | 3 | 4
Not completed — Investigator's discretion | 1 | 2
Not completed — Withdrew consent | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized into the study and received at least 1 dose of study drug.
Groups:
- B/F/TAF: Double-Blind Phase: B/F/TAF 50/200/25 mg FDC tablet + ABC/DTG/3TC placebo orally once daily for at least 48 weeks, without regard to food.
  OL Extension Phase: After Week 48, participants in a country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
- Total: Total of all reporting groups
Arm/Group | B/F/TAF | ABC/DTG/3TC | Total
Number analyzed (Participants) | 282 | 281 | 563
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11.1) | 45 (11.5) | 45 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 29 | 64
  Male | 247 | 252 | 499
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information.
  Participants
    American Indian or Alaska Native | 2 | 2 | 4
    Asian | 9 | 9 | 18
    Black | 59 | 62 | 121
    Native Hawaiian or Pacific Islander | 3 | 0 | 3
    White | 206 | 202 | 408
    Other | 3 | 3 | 6
    Not Permitted | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information
  Participants
    Hispanic or Latino | 46 | 52 | 98
    Not Hispanic or Latino | 236 | 227 | 463
    Not Permitted | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 13 | 22 | 35
  Belgium | 1 | 1 | 2
  United States | 203 | 198 | 401
  Italy | 1 | 1 | 2
  United Kingdom | 3 | 3 | 6
  France | 4 | 8 | 12
  Germany | 17 | 11 | 28
  Spain | 31 | 31 | 62
  Australia | 9 | 6 | 15
HIV-1 RNA Categories [Count of Participants; unit: Participants]
  < 50 copies/mL | 278 | 272 | 550
  ≥ 50 copies/mL | 4 | 9 | 13
CD4 Cell Count [Mean (Standard Deviation); unit: cell/µL] | 752 (302.2) | 694 (291.6) | 723 (298.1)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  ≥ 50 to < 200 cells/μL | 6 | 4 | 10
  ≥ 200 to < 350 cells/μL | 16 | 30 | 46
  ≥ 350 to < 500 cells/μL | 33 | 42 | 75
  ≥ 500 cells/μL | 227 | 205 | 432

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Virologic Failure (HIV-1 RNA ≥ 50 Copies/mL) as Defined by the Modified US FDA-defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA ≥ 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: The Full Analysis Set included participants who were randomized into the study and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 282 | 281
percentage of participants | 1.1 | 0.4
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Non-Inferiority — A sample size of 260 participants per treatment group would provide at least 90% power to detect a noninferiority margin of 4% in difference in percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Wk 48, between B/F/TAF group and ABC/DTG/3TC group. Sample size was based on assumptions that both treatment groups have 2% of participants with HIV-1 RNA ≥ 50 copies/mL at Wk 48 and that the non-inferiority margin is 4%, and that the significance level of the test is at a one-sided 0.025 level; Difference in Percentages = 0.7, 95.002% CI 2-sided [-1.0 to 2.8] — The differences in percentages of participants between treatment groups and their 95.002% CIs were calculated based on an unconditional exact method using 2 inverted 1-sided tests
Statistical Analysis 2: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Superiority; p = 0.62, Fisher Exact

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL as Defined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 282 | 281
percentage of participants | 93.6 | 95.0
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Non-Inferiority — It would be concluded that B/F/TAF is noninferior to ABC/DTG/3TC if the lower bound of the 2-sided 95.002% CI of the difference between treatment groups (B/F/TAF group -ABC/DTG/3TC group) in the percentage of participants with HIV-1 RNA < 50 copies/mL is greater than -10%; Difference in Percentages = -1.4, 95.002% CI 2-sided [-5.5 to 2.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Superiority; p = .59, Fisher Exact

3. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 265 | 267
cells/µL | -31 (181.3) | 4 (191.0)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.031, ANOVA; Difference in least squares means = -35, 95% CI 2-sided [-67 to -3]

4. Secondary Outcome: Spine Bone Mineral Density (BMD) at Baseline
Time Frame: Baseline
Population: The Spine dual X-ray absorptiometry (DXA) analysis Set included participants who were randomized into the study, received at least 1 dose of study drug, and had nonmissing baseline spine BMD values.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 256 | 262
g/cm^2 | 1.124 (0.1833) | 1.103 (0.1548)

5. Secondary Outcome: Percentage Change From Baseline in Spine BMD at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 233 | 244
percentage change | 0.692 (3.1296) | 0.416 (2.9973)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.33, ANOVA; Difference in least squares means = 0.276, 95% CI 2-sided [-0.275 to 0.827]

6. Secondary Outcome: Hip Bone Mineral Density at Baseline
Time Frame: Baseline
Population: The Hip DXA Analysis Set included participants who were randomized into the study, received at least 1 dose of study drug, and had nonmissing baseline hip BMD values.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 256 | 265
g/cm^2 | 1.006 (0.1471) | 0.996 (0.1363)

7. Secondary Outcome: Percentage Change From Baseline in Hip BMD at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | B/F/TAF | ABC/DTG/3TC
Number analyzed (Participants) | 229 | 242
percentage change | 0.156 (2.2138) | 0.299 (2.1077)
Statistical Analysis 1: Comparison: B/F/TAF vs ABC/DTG/3TC; Test type: Other; p = 0.47, ANOVA; Difference in least squares means = -0.143, 95% CI 2-sided [-0.534 to 0.248]

ADVERSE EVENTS:
Time Frame: First dose date up to 169 weeks plus 30 days
Description: The Safety Analysis Set included participants who were randomized into the study and received at least 1 dose of study drug.
Groups:
- Double-Blind: B/F/TAF: B/F/TAF (50/200/25 mg) FDC tablet + ABC/DTG/3TC placebo orally once daily for at least 48 weeks, without regard to food.
- Double-Blind: ABC/DTG/3TC: ABC/DTG/3TC (600/50/300 mg) FDC tablet + B/F/TAF placebo orally once daily for at least 48 weeks, without regard to food.
- Open-label Extension: B/F/TAF From B/F/TAF: Participants who received B/F/TAF in double-blind phase and from country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
- Open-label Extension: B/F/TAF From ABC/DTG/3TC: Participants who received ABC/DTG/3TC in double-blind phase and from country where B/F/TAF was not available were given the option to receive B/F/TAF orally once daily for up to 96 weeks in the open-label extension phase.
Arm/Group | Double-Blind: B/F/TAF | Double-Blind: ABC/DTG/3TC | Open-label Extension: B/F/TAF From B/F/TAF | Open-label Extension: B/F/TAF From ABC/DTG/3TC
All-Cause Mortality (participants affected / at risk) | 2/282 | 0/281 | 1/259 | 1/265
Serious Adverse Events (participants affected / at risk) | 17/282 | 26/281 | 24/259 | 11/265
Other Adverse Events (participants affected / at risk) | 122/282 | 132/281 | 84/259 | 82/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind: B/F/TAF (N=282) | Double-Blind: ABC/DTG/3TC (N=281) | Open-label Extension: B/F/TAF From B/F/TAF (N=259) | Open-label Extension: B/F/TAF From ABC/DTG/3TC (N=265)
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial bridging (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Macular detachment (Eye disorders) | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 2 | 0 | 1
Acute hepatitis C (Infections and infestations) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1 | 0
Eye infection syphilitic (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Large intestine infection (Infections and infestations) | 1 | 1 | 0 | 0
Lymphadenitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Shigella infection (Infections and infestations) | 0 | 1 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Testicular seminoma (pure) stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Hemiplegic migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0
Self-injurious ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Substance abuse (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind: B/F/TAF (N=282) | Double-Blind: ABC/DTG/3TC (N=281) | Open-label Extension: B/F/TAF From B/F/TAF (N=259) | Open-label Extension: B/F/TAF From ABC/DTG/3TC (N=265)
Diarrhoea (Gastrointestinal disorders) | 26 | 18 | 20 | 11
Nausea (Gastrointestinal disorders) | 6 | 16 | 3 | 1
Bronchitis (Infections and infestations) | 11 | 15 | 11 | 8
Nasopharyngitis (Infections and infestations) | 21 | 22 | 20 | 22
Sinusitis (Infections and infestations) | 11 | 15 | 9 | 13
Upper respiratory tract infection (Infections and infestations) | 34 | 32 | 22 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 18 | 8 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 13 | 13 | 6
Headache (Nervous system disorders) | 19 | 23 | 5 | 9
Insomnia (Psychiatric disorders) | 9 | 22 | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Original (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT02603120/Prot_004.pdf
  • Study Protocol: Amendment 2 (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT02603120/Prot_006.pdf
  • Study Protocol: Amendment 1 (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT02603120/Prot_007.pdf
  • Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT02603120/SAP_008.pdf